CLINICAL TRIAL: NCT03718013
Title: Efficacy and Safety of Accelerated Transcranial Magnetic Stimulation With H1-coil (dTMS); Randomized Controlled Equivalence Trial
Brief Title: Efficacy and Safety of Accelerated Transcranial Magnetic Stimulation With H1-coil (dTMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sveti Ivan Psychiatric Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: acceleratedDTMS
Record Dates: First submitted 2018-10-16; First posted 2018-10-24 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- accelerated dTMS (Experimental)
  Interventions: Device: accelerated deep TMS
- standard dTMS (Active Comparator)
  Interventions: Device: standard deep TMS

INTERVENTIONS:
Device: accelerated deep TMS — subjects treated with deep TMS twice a day (6-8 hours between two applications), during 2 weeks
  Arms: accelerated dTMS
Device: standard deep TMS — standard deep TMS treatment: once a day, during 4 weeks
  Arms: standard dTMS

SUMMARY:
The purpose of this study is to examine the efficacy and safety of accelerated transcranial magnetic stimulation with H1-coil (deep TMS) for treatment of patients diagnosed with major depressive disorder (MDD). Subjects will be randomized into two groups: experimental (treated with accelerated deep TMS: twice a day (6-8 hours between two applications), during 2 weeks) and control group (standard deep TMS treatment: once a day, during 4 weeks). Participants and designated clinicians will complete a battery of instruments that measure relevant symptoms (HAM-D17 and BDI-II scales), global functioning (CGI and PHQ-9 scales), quality of life (EQ-5D-5L questionnaire), and cognitive functions (MoCA test). Measurements will be done in 4 time points: after the inclusion, after the first week of treatment, after the second week (the end of treatment for experimental group), after the fourth week (the end of treatment for control group), and after 1 month (follow-up for both groups). Interim data analysis is planned at the time when at least 30 participants are involved in both groups. Patients whose baseline score on HAM-D17 is equal or greater than 24 (very severe depression) will be included in another study; they will be treated with accelerated deep TMS twice a day during 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed major depressive disorder (ICD10: F32.1, F32.2, F33.1, F33.2)
* current depressive episode lasts for at least 4 weeks
* HAM-D17 score ≥15
* CGI-Score ≥4
* inadequate response to antidepressant therapy

Exclusion Criteria:

* diagnosed psychotic disorder
* diagnosed depressive disorder with psychotic features
* diagnosed bipolar affective disorder
* diagnosed posttraumatic stress disorder
* diagnosed obsessive-compulsive disorder
* anxiety disorder or personality disorder as primary diagnoses
* alcohol or drug addiction
* neurological disorders and brain implants
* pregnancy
* former TMS treatment within 6 months
* unable to complete the questionnaires

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage improvement in the Hamilton Rating Scale for Depression (HAM-D) scores | 8 weeks
  The Hamilton Rating Scale for Depression (HAM-D) is a clinician-administered depression assessment scale. The original version contains 17 items pertaining to symptoms of depression experienced over the past week. The items are scored either on a 3-point or 5-point scale, and all the values are summed to obtain a total scale score. Scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression and scores over 24 are indicative of severe depression (the maximum score being 52).

SECONDARY OUTCOMES:
Treatment response | 8 weeks
  ≥50% decrease in scores on the Hamilton Rating Scale for Depression (HAM-D)
The proportion of patients who experienced complete remission of the disease | 8 weeks
Percentage improvement in BDI-II scores | 8 weeks
  The Beck Depression Inventory (BDI-II) is a 21-question multiple-choice self-report inventory for measuring the severity of depression. Each answer is scored on a scale value of 0 to 3. All the values are summed to obtain a total scale score. Higher total scores indicate more severe depressive symptoms. Scores of 0-13 are considered as minimal depression,14-19 suggest mild depression, 20-28 moderate depression, and 29-63 severe depression.
Change in perceived quality of life (EQ-5D-5L scale) | 8 weeks
  The EQ-5D-5L is a standardised self-report measure of health status developed by the EuroQol Group. It consists of the descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises the 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression), and each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent´s decision results in a 1-digit number expressing the level selected for that dimension. The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' (number 100) and 'the worst health you can imagine' (number 0). The respondents are asked to mark an X on the scale to indicate how their health is today and then to write the number they marked on the scale in the box below.
Change in cognitive functions (MoCA test) | 8 weeks
  The Montreal Cognitive Assessment (MoCA) is a one-page 30-point screening assessment for detecting cognitive impairment. It assesses several cognitive domains: the short-term memory recall task (5 points), visuospatial abilities (4 points), multiple aspects of executive functions (4 points), attention, concentration, and working memory (6 points), language (5 points), and orientation to time and place (6 points). A score of 26 or over is considered to be normal.

CONTACTS AND LOCATIONS:
Locations (1):
- PB Sveti Ivan, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided